CLINICAL TRIAL: NCT00006307
Title: Epidemiology of Body Mass Index Rebound
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 915; R01HL064022 (NIH)
Record Dates: First submitted 2000-09-28; First posted 2000-09-29 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2008-01

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Obesity

SUMMARY:
To investigate the relationship between obesity, body mass index (BMI) rebound, body composition changes, associated factors (e.g., diet, physical activity), and cardiovascular risk factor status in a longitudinal study of young children, age three at the beginning of the study.

DETAILED DESCRIPTION:
BACKGROUND:

Obesity is the most prevalent nutritional problem in the United States. It appears that both the prevalence and severity of obesity have been increasing in recent years. Obesity often begins in childhood and has a number of severe sequelae, including non insulin dependent diabetes mellitus and cardiovascular disease. Unfortunately, obesity is very resistant to treatment. This places a premium on prevention. However, the identification of clinically useful predictors of obesity which are present prior to the onset of excess weight gain has been problematic. Recently, it has been shown that the timing of body mass index (BMI) rebound may be a predictor of future obesity. BMI increases during the first year of life. It then declines until it reaches a minimum value during childhood and subsequently increases into adolescence and adulthood. The nadir of BMI is called BMI rebound. Studies have shown that BMI rebound at a young age is associated with increased risk of obesity later in life. Currently, very little is known about the epidemiology of BMI rebound.

DESIGN NARRATIVE:

The investigation is a cohort study designed to follow 320 children from age three to age seven years. The study design will be a longitudinal one in which the children will be followed for a period of four years during which repeat measurements of body composition, diet, and physical activity will be made every four months. Parental height and weight data will be collected, in addition to family health history, parental smoking and alcohol intake.

ELIGIBILITY:
No eligibility criteria

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2000-08; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Daniels — Children's Hospital & Medical Center

REFERENCES:
- [Background] Burdette HL, Whitaker RC, Daniels SR. Parental report of outdoor playtime as a measure of physical activity in preschool-aged children. Arch Pediatr Adolesc Med. 2004 Apr;158(4):353-7. doi: 10.1001/archpedi.158.4.353. PMID 15066875